CLINICAL TRIAL: NCT05100368
Title: The Prognostic Value of Serum Biomarkers in Ewing's Sarcoma
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: PROSARC
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-03

CONDITIONS: Sarcoma, Ewing
Keywords: sarcoma; ewing
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with Ewing's Sarcoma and osteosarcoma with established diagnosis
  Interventions: Other: patients

INTERVENTIONS:
Other: patients — Patients with Ewing's Sarcoma and osteosarcoma with established diagnosis

SUMMARY:
Extraction of laboratory data from blood tests prior to surgical and chemotherapy and other histological, clinical and instrumental data related to the patient's history from the digitized medical Digitized medical records and analysis of the same. The medical records of 1000 patients from January 1, 2000, until December 31, 2020

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ewing's Sarcoma and osteosarcoma with established diagnosis;
* Patients with age ≥ 2 years;
* Minimum follow-up duration of 2 years;
* Medical records, complete blood work and instrumental examinations; Regular follow-up.

Exclusion Criteria:

* Patients with Ewing's sarcoma or osteosarcoma who have received medical treatment (surgery radiotherapy or chemotherapy) in other institutions prior to admission to the Rizzoli Orthopaedic Institute.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Ewing's sarcoma or osteosarcoma
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
5-year survival | at baseline (Day0)
  Evaluation of 5-year survival in relation to histologic, laboratory, clinical, and instrumental laboratory, clinical and instrumental factors

SECONDARY OUTCOMES:
Rate of local recurrence | at baseline (Day0)
  Evaluation of the rate of local recurrence and distant metastasis in relation to prognostic factors histological, laboratory, clinical and instrumental factors;

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakamura T, Grimer RJ, Gaston CL, Watanuki M, Sudo A, Jeys L. The prognostic value of the serum level of C-reactive protein for the survival of patients with a primary sarcoma of bone. Bone Joint J. 2013 Mar;95-B(3):411-8. doi: 10.1302/0301-620X.95B3.30344. PMID 23450030
- [Result] Li YJ, Yang X, Zhang WB, Yi C, Wang F, Li P. Clinical implications of six inflammatory biomarkers as prognostic indicators in Ewing sarcoma. Cancer Manag Res. 2017 Sep 28;9:443-451. doi: 10.2147/CMAR.S146827. eCollection 2017. PMID 29033609
- [Result] Aggerholm-Pedersen N, Maretty-Kongstad K, Keller J, Baerentzen S, Safwat A. The Prognostic Value of Serum Biomarkers in Localized Bone Sarcoma. Transl Oncol. 2016 Aug;9(4):322-8. doi: 10.1016/j.tranon.2016.05.006. PMID 27567955